CLINICAL TRIAL: NCT03686111
Title: NUCLEAR LAMINA, OVARIAN AGE AND MEDICAL ASSISTANCE TO PROCREATION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-03; 2017-A01258-45 (Other: ANSM)
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- infertile patientes with medical assistance to procreation
  Interventions: Diagnostic Test: oocytes collect
- Infertile patientes with induction of ovulation to give their
  Interventions: Diagnostic Test: oocytes collect

INTERVENTIONS:
Diagnostic Test: oocytes collect — After stimulation, an echo-guided oocyte puncture is performed under anesthesia

SUMMARY:
The nuclear lamina (LN) consists of a network of proteins interposed between the chromatin and the internal nucleic membrane, to which it is closely associated. LN consists essentially of lamins encoded by the LMNA (Lamines A / C), LMNB1 and LMNB2 genes (BI, B2, B3 lamins). Malfunctions of the A / C-type laminates causing the production of a toxic isoform called progerin are directly responsible for various serious pathologies such as Progeria Hutchingson-Gilford. This rare disease is characterized by accelerated pathological aging. Moreover, it is known that progerin is produced in the absence of any mutation of the gene LMNA is involved in the physiological aging of tissus.

The ovarian reserve of a woman is a parameter that changes with age. Although this progressive loss is inevitable in the course of life, the kinetics of this ovarian exhaustion appear variable according to the women, sometimes leading to an accelerated loss causing a discordance between the female age and the ovarian age. But ovarian age becomes a major prognostic parameter to be taken into account during any attempt at medical assistance to procreation (AMP) and is often incriminated in the failures of MPAs. There are currently few markers to predict the quality of ovarian response of women to ovarian stimulation, let alone the quality of the oocytes retrieved. However, their quality directly influences their ability to give an evolving embryo and therefore a pregnancy Our team has previously shown that type B laminates are involved in human spermiogenesis, and highlighted the human B3 isoform. These very encouraging results obtained on human spermatogenesis, have prompted us to also look at the potential interest of the exploration of the nuclear lamina within the human ovary.

The aim of this project is therefore to continue the exploration of the nuclear lamina and its potential role on the quality of human gametes, by studying the follicular ovarian cells surrounding the oocyte. These cells express A / C type lamins and sometime progerin Investigators want to conduct a prospective pilot study in a cohort of 40 women in MPA, aged between 20 and 42 years. The main objective is to compare the levels of expression of the A / C, B and progerin laminae in the follicular cells of 2 groups of women: a group of infertile patients managed to induce ovulation in order to Intraconjugal AMP and a group of women managed to induce ovulation to give their oocytes. For this purpose, investigators will analyze the expression of the A / C and B lamins in RT-PCR, the localization of the lamins and progerin in immunofluorescence, and will look for quantitative variations in the production of A / C and / or progerin lamins by western- blot, depending on the age of the patients.

This pilot study will allow investigators to characterize for the first time the LN of human follicular cells. They should highlight variations in the expression and / or localization of lamins and possibly progerin in patients tested according to their age and / or ovarian reserve. The team preliminary results showed that this track deserves to be explored. This is an excellent opportunity to bring new insights into the understanding of the mechanisms responsible for alteration of ovarian reserve in women and the prognosis of MPA attempts.

Finally, this approach could serve as a basis for a larger, multicenter study. These markers could represent new diagnostic markers to be taken into account to evaluate the chances of pregnancy of each woman in AMP.

ELIGIBILITY:
Inclusion Criteria:

* Patientes going through induction of ovulation by dual-triggering antagonist protocol
* Body mass index<30

Exclusion Criteria:

* Patientes going through induction of ovulation for fertility conservation because of cancer treatment initiation.

Ages: 20 Years to 42 Years | Sex: Female
Age Groups: Adult
Study Population: Patients recruited will be either women managed for in vitro fertilization with micro injection type, or donor eggs stimulated to obtain oocytes used for in vitro micro-injection fertilization.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
percent of expression progerin in follicular cells | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Emilie GARRIDO, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France